CLINICAL TRIAL: NCT00345085
Title: Comparison of Higher Order Aberrations and Contrast Sensitivity Between Acrysof SN60AT, SN60WF and Restore Intraocular Lenses
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: James P. McCulley, MD, UTSW Medical Center at Dallas
Other Study IDs: 052006-029
Record Dates: First submitted 2006-06-23; First posted 2006-06-27 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2008-06

CONDITIONS: Refractive Errors
MeSH Terms: conditions — Refractive Errors | interventions — Contrast Sensitivity

INTERVENTIONS:
Device: Wavefront and Contrast Sensitivity

SUMMARY:
This project involves evaluation of post operative contrast sensitivity and wavefront aberration results among patients implanted with standard monofocal lenses (Acrysof SN60AT/SN60WF) and the new presbyopic correcting multifocal lens (Acrysof ReSTOR). Higher Order aberrations are visual phenomena such as glare and haloes. They are more prevalent after cataract surgery and can affect night driving.

DETAILED DESCRIPTION:
The Project involves evaluation of contrast sensitivity and higher order aberrations in patients implanted with SN60AT, SN60WF and ReSTOR intraocular lenses. Patients in the department of Ophthalmology will be asked to participate in the study on a routine postoperative visit at least 3 months after cataract surgery. Patients will be asked to sign a consent form prior to participation. Wavefront analysis involves the patient resting their chin in a device similar to a slit lamp; they focus on a distant light and the machine performs the measurements in mesopic and scotopic conditions (light and dark). Contrast sensitivity is a measure of how faded or washed out an image can be before it becomes indistinguishable from a uniform field; it involves the patient identifying patterns on a chart. Wavefront analysis and contrast sensitivity are noninvasive tests that do not employ sedation or anesthesia and does not expose the patient to x-rays or microwaves. The proposed research will not alter usual standard postoperative care and can be done on a routine office visit.

ELIGIBILITY:
Inclusion Criteria: All subject implanted with either SN60AT, SN60WF or ReSTOR intraocular lenses after cataract removal. Subjects include those 18 yrs and over, male and female, all races. Patients will sign an informed consent

Exclusion Criteria: Patients younger than 18 yrs. Patients with other concurrent visually significant ophthalmic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-03; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
post operative wavefront aberration

SECONDARY OUTCOMES:
post operative contrast sensitivity

CONTACTS AND LOCATIONS:
Overall Officials: James P McCulley, M.D., Study Chair — UTSW Medical Center at Dallas; Shady Awwad, M.D., Principal Investigator — UTSW Medical Center at Dallas
Locations (1):
- UTSW Medical Center at Dallas, Dallas, Texas, United States